CLINICAL TRIAL: NCT04214860
Title: Phase I Study of APR-246 in Combination With Venetoclax and Azacitidine in TP53-Mutant Myeloid Malignancies
Brief Title: APR-246 in Combination With Venetoclax and Azacitidine in TP53-Mutant Myeloid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aprea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A19-11184
Record Dates: First submitted 2019-12-12; First posted 2020-01-02 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Myeloid Malignancy
MeSH Terms: interventions — eprenetapopt; venetoclax; Azacitidine

STUDY DESIGN:
Intervention Model Description: The study will include a safety lead-in dose-finding portion followed by the expansion portion. During the safety lead-in portion of the study, two cohorts will independently enroll patients following a 3 + 3 design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APR-246 (Experimental): APR-246 4.5 g/day
  Interventions: Drug: APR-246; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: APR-246 — APR-246 4.5 g/day
Drug: Venetoclax — Venetoclax 400 mg once daily
Drug: Azacitidine — Subcutaneous injection, or intravenous infusion

SUMMARY:
This clinical trial is a Phase I, open-label, dose-finding and cohort expansion study to determine the safety and preliminary efficacy of APR-246 in combination with venetoclax and azacitidine in patients with myeloid malignancies.

DETAILED DESCRIPTION:
This study will enroll adult male and female patients of age ≥ 18 years with documented diagnosis of AML, according to WHO classification, and documented TP53 mutation which is not benign or likely benign, who also meet the eligibility requirements of this protocol.

The study will include a safety lead-in dose-finding portion followed by expansion portion. During the safety lead-in portion of the study, two cohorts will independently enroll patients following a 3 + 3 design. Each cohort will enroll up to 6 patients.

The expansion portion will begin once the recommended phase II dose (RP2D) of APR-246 in combination with venetoclax and in combination with venetoclax and azacitidine have been determined in order to assess the antitumor activity of these combinations.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent and ability to comply with protocol requirements.
2. Documented diagnosis of AML according to World Health Organization WHO) classification
3. Adequate organ function as defined by the following laboratory values:

   1. Creatinine clearance > 30 mL/min
   2. Total serum bilirubin < 1.5 × ULN
   3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 × ULN
4. Age ≥18 years
5. At least one TP53 mutation
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
7. Projected life expectancy of ≥ 12 weeks.
8. Negative serum or urine pregnancy test
9. Females of childbearing potential and males with female partners of childbearing potential must be willing to use an effective form of contraception

Exclusion Criteria:

1. Prior treatment for TP53-mutant AML (*dependent upon treatment arm assigned).
2. Known history of HIV or active hepatitis B or active hepatitis C infection.
3. Any of the following cardiac abnormalities:

   1. Myocardial infarction within six months prior to registration;
   2. New York Heart Association Class III or IV heart failure or known left ventricular ejection fraction (LVEF) < 40%;
   3. A history of familial long QT syndrome;
   4. Symptomatic atrial or ventricular arrhythmias
   5. QTcF ≥ 470 msec, unless due to underlying bundle branch block and/or pacemaker and with approval of the medical monitor.
4. Concomitant malignancies for which patients are receiving active therapy
5. Known active CNS involvement from AML.
6. Malabsorption syndrome
7. Pregnancy or lactation.
8. Active uncontrolled systemic infection (viral, bacterial or fungal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt CC, Tampa, Florida
  - Northwestern Medicine, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Cancer Center, New York, New York
  - Memorial Sloan Kettering CC, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia-Manero G, Goldberg AD, Winer ES, Altman JK, Fathi AT, Odenike O, Roboz GJ, Sweet K, Miller C, Wennborg A, Hickman DK, Kanagal-Shamanna R, Kantarjian H, Lancet J, Komrokji R, Attar EC, Sallman DA. Eprenetapopt combined with venetoclax and azacitidine in TP53-mutated acute myeloid leukaemia: a phase 1, dose-finding and expansion study. Lancet Haematol. 2023 Apr;10(4):e272-e283. doi: 10.1016/S2352-3026(22)00403-3. PMID 36990622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cohort 2 APR-246 + VEN + AZA Safey Lead-In and Expansion data was combined for reporting purposes.
Groups:
- Cohort 1: APR-246 4.5 g/day
  APR-246: APR-246 4.5 g/day day 1-4
  Venetoclax: Venetoclax 400 mg once daily days 1-28
  Safety Lead-In
- Cohort 2: PR-246 4.5 g/day
  APR-246: APR-246 4.5 g/day day 1-4
  Venetoclax: Venetoclax 400 mg once daily days 1-28
  Azacitidine: Azacitidine 75 mg/m² on days 1-7.
  Safety Lead-In + Expansion
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 6 | 45
Completed | 6 | 43
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: APR-246 4.5 g/day
  APR-246: APR-246 4.5 g/day
  Venetoclax: Venetoclax 400 mg once daily
- Cohort 2: APR-246 4.5 g/day
  APR-246: APR-246 4.5 g/day
  Venetoclax: Venetoclax 400 mg once daily
  Azacitidine: Subcutaneous injection, or intravenous infusion
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 6 | 43 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 16 | 18
  >=65 years | 4 | 27 | 31
Age, Continuous [Median (Full Range); unit: years] | 69 [45 to 76] | 67 [27 to 81] | 67 [27 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 20 | 24
  Male | 2 | 23 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 3 | 37 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 43 | 49

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Tolerabililty and the Incidence of Treatment-Emergent Adverse Events of Administration of APR 246 in Combination With Venetoclax and Azacitidine in Patients With TP53 Mutant Myeloid Malignancies.
Description: 1. Dose-limiting toxicities (DLTs), classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 5.0).
Time Frame: From baseline until event occures, i.e. through study completion, an average of 1 year
Measure: Number; unit: DLTs
Groups:
- Cohort 1: APR-246 4.5 g/day
  APR-246: APR-246 4.5 g/day day 1-4
  Venetoclax: Venetoclax 400 mg once daily days 1-28
- Cohort 2: PR-246 4.5 g/day
  APR-246: APR-246 4.5 g/day day 1-4
  Venetoclax: Venetoclax 400 mg once daily days 1-28
  Azacitidine: Azacitidine 75 mg/m² on days 1-7.
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 43
DLTs | 0 | 0

2. Primary Outcome: To Evaluate the Tolerabililty and the Incidence of Treatment-Emergent Adverse Events of Administration of APR 246 in Combination With Venetoclax and Azacitidine in Patients With TP53 Mutant Myeloid Malignancies.
Description: 2. Frequency of treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs) related to APR-246 in combination with venetoclax and azacitidine during the trial.
Time Frame: From baseline until event occures, i.e. through study completion, an average of 1 year
Population: Any Serious TEAEs
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 43
Participants | 5 | 32

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 6/6 | 26/43
Serious Adverse Events (participants affected / at risk) | 5/6 | 32/43
Other Adverse Events (participants affected / at risk) | 6/6 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=43)
Pneumonia (Infections and infestations) | 0 | 6
Sepsis (Infections and infestations) | 2 | 4
Diverticulitis (Infections and infestations) | 0 | 2
abdominal abscess (Infections and infestations) | 0 | 1
Bacteremia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 1
Infusion Site Infection (Infections and infestations) | 0 | 1
Periorbital Celluitis (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Sinusitis Fungal Infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 13
Anemia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Obstruction Gastric (Gastrointestinal disorders) | 0 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 1
Mucosal Inflammation (General disorders) | 1 | 1
Death (General disorders) | 0 | 1
Gait Disturbance (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Tachycaridia (Cardiac disorders) | 1 | 0
Acute Respiratory distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkelaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Hemorrahge intracranial (Nervous system disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Subdural Harmatoma (Injury, poisoning and procedural complications) | 0 | 2
Blood Creatinine Increased (Investigations) | 0 | 1
Blood bilirubin Increased (Investigations) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cytokine release syndorme (Immune system disorders) | 0 | 1
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute Febrile Neutrophilic Deramotsis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6) | Cohort 2 (N=43)
Nasuea (Gastrointestinal disorders) | 6 | 27
Diarrhea (Gastrointestinal disorders) | 3 | 24
Vomiting (Gastrointestinal disorders) | 3 | 20
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 19
Decreased Appetite (Gastrointestinal disorders) | 2 | 18
Constipation (Gastrointestinal disorders) | 3 | 15
Hypokalemia (Metabolism and nutrition disorders) | 3 | 14
Platelet Count Decreased (Investigations) | 2 | 14
Dizziness (Nervous system disorders) | 3 | 13
Edema Peripheral (General disorders) | 3 | 13
Hypotension (Vascular disorders) | 2 | 13
Anemia (Blood and lymphatic system disorders) | 1 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Fatgiue (General disorders) | 2 | 11
White Blood Cell Count Deceased (Investigations) | 0 | 12
Pneumonia (Infections and infestations) | 2 | 10
Headache (Nervous system disorders) | 3 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 9
chills (General disorders) | 1 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Neutrophil count decreased (Investigations) | 2 | 8
tremor (Nervous system disorders) | 2 | 8
Confusional State (Psychiatric disorders) | 1 | 8
Sinus Tachycardia (Cardiac disorders) | 1 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 7
Insomnia (Psychiatric disorders) | 3 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 8
contusion (Skin and subcutaneous tissue disorders) | 2 | 6
Hyperphospataemia (Metabolism and nutrition disorders) | 2 | 6
Abdominal Distension (Gastrointestinal disorders) | 0 | 7
Dysgeusia (Gastrointestinal disorders) | 0 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 7
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3 | 5
Abdominal Pain (Gastrointestinal disorders) | 1 | 6
Gait Disturbance (General disorders) | 1 | 6
Rhinorrhoea (Infections and infestations) | 1 | 6
Sepsis (Infections and infestations) | 2 | 5
Stomatitis (Gastrointestinal disorders) | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6
Pyrexia (General disorders) | 3 | 4
Electrocardiogram QT prolonged (Cardiac disorders) | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dysuria (Renal and urinary disorders) | 0 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pain (General disorders) | 0 | 5
Pain in extremity (General disorders) | 0 | 5
Asthenia (Musculoskeletal and connective tissue disorders) | 1 | 4
Injection site reaction (General disorders) | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT04214860/Prot_SAP_000.pdf